CLINICAL TRIAL: NCT06973382
Title: Intervention Study of a Comprehensive Pulmonary Rehabilitation Program on Quality of Life and Prognosis in Patients With Pulmonary Arterial Hypertension
Brief Title: Effects of Pulmonary Rehabilitation on Quality of Life and Health in Pulmonary Arterial Hypertension Patients
Acronym: EPRQoL-PAH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Beijing Municipal Health Commission (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-KE-62-1
Record Dates: First submitted 2025-05-14; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-02

CONDITIONS: PAH; CTEPH

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Pulmonary Rehabilitation Program (Experimental)
  Interventions: Behavioral: Comprehensive Pulmonary Rehabilitation Program
- Standard Pulmonary Rehabilitation (Active Comparator)
  Interventions: Behavioral: Standard Pulmonary Rehabilitation

INTERVENTIONS:
Behavioral: Comprehensive Pulmonary Rehabilitation Program — Combined Aerobic + Resistance Training Program Mode: Cycle ergometry (stationary bicycle) Frequency: 3-5 sessions per week Program Duration: 12 weeks
  Session Structure:
  * 5-minute warm-up
  * Continuous or interval training (15-30 minutes)
  * 5-minute cool-downesistance Exercise Component
  Mode: Dumbbell exercises + cycle ergometry
  Frequency: 3 sessions per week
  Program Duration: 12 weeks
  Session Structure:
  * 5-minute warm-up
  * Training session (10-20 minutes)
  * 5-minute cool-down
  Arms: Comprehensive Pulmonary Rehabilitation Program
Behavioral: Standard Pulmonary Rehabilitation — xercise Components:
  Aerobic Exercise
  Mode: Walking or jogging
  Resistance Exercise
  Mode: Elastic bands or dumbbells
  Training Parameters:
  Session Duration: ≥35 minutes (combined aerobic + resistance)
  Frequency: 3-5 sessions per week
  Program Duration: 12 weeks
  Arms: Standard Pulmonary Rehabilitation

SUMMARY:
Pulmonary hypertension (PH) is a major global health concern, affecting approximately 1% of the world's population. With global aging and increased life expectancy, its incidence continues to rise. PH is a progressive and disabling disease, with studies showing its progression correlates with worsening symptoms and increased mortality. Even with targeted medications, the prognosis remains poor across PH subtypes, with PAH patients showing only a 49% 7-year survival rate. The 2022 ESC/ERS guidelines emphasize that PH management requires a comprehensive, multidisciplinary approach. Beyond pharmacological and surgical treatments, rehabilitation has demonstrated benefits in improving exercise capacity, quality of life, functional class, and peak oxygen consumption. However, research on specific and effective comprehensive pulmonary rehabilitation programs remains lacking.

ELIGIBILITY:
Inclusion Criteria:Confirmed PH Diagnosis:

Right heart catheterization-confirmed pulmonary hypertension

Meets 2022 ESC/ERS Guidelines diagnostic criteria for:

* Group 1 (PAH) or
* Group 4 (CTEPH/other pulmonary artery obstructions)

Stabilized Treatment Status:

Group 1 (PAH): Received ≥3 months of targeted drug therapy

Group 4 (CTEPH): Completed ≥6 sessions of BPA* or reached therapeutic endpoint

Functional Capacity:

WHO Functional Class I-III

Age: ≥18 years

Consent: Willing to provide written informed consent -

Exclusion Criteria:Physical Limitations:

Unable to perform pulmonary rehabilitation exercises due to disability or congenital malformations

Cardiopulmonary Testing Contraindications:

Medically unfit to complete CPET (cardiopulmonary exercise testing) after evaluation

Poor Compliance:

History of non-adherence making protocol completion unlikely

Life Expectancy:

Prognosis ≤1 year

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
6MWD | 12week

IPD SHARING:
Plan to Share IPD: No